CLINICAL TRIAL: NCT01516294
Title: A Pilot, Single-center, Interventional Clinical Trial in Which Subjects With Polypoidal Choroidal Vasculopathy (PCV) Secondary to Age-Related Macular Degeneration (AMD) Will Receive Low Voltage Stereotactic Radiotherapy (IRay®) Treatment and Lucentis® Treatment as Needed.
Brief Title: IRay to Treat Polypoidal Choroidal Vasculopathy (PCV) Secondary to Age-Related Macular Degeneration (AMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oraya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLH004
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Polypoidal Chorodial Vasculopathy; Age Related Macular Degeneration
Keywords: AMD; PCV; Iray; radiation; retina; macula; radiotherapy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iray plus Lucentis (Experimental): open label arm in which all subjects recieve a single 16 gy dose of radiation plus an injection of Lucentis.
  Interventions: Radiation: Iray

INTERVENTIONS:
Radiation: Iray — The Oraya IRay stereotactic radiotherapy device will be used to deliver a 16 Gy dose of radiation to the macula. The radiotherapy will be delivered in a single session utilizing three sequential beams, each depositing 5.3 Gy at the macula through calculated scleral entry points, crossing the pars plana region of the eye, and overlapping at the same region of the macula.

SUMMARY:
This study will evaluate the efficacy of IRay treatment in patients with Polypoidal Choroidal Vasculopathy (PCV)secondary to AMD as determined by the change in the proportion of lesion activity and lesion size at 12 months.

DETAILED DESCRIPTION:
This is a single-center, interventional clinical trial in which subjects will receive 16 Gy of IRay treatment and Lucentis, followed by Lucentis treatment as needed to evaluate the efficacy of IRay treatment in patients with PCV as determined by the change in the proportion of lesion activity and lesion size at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCV, naïve or previously treated with Lucentis injections and Photodynamic therapy (PDT) using Visudyne.
* Must have a total lesion size of <12 disc areas and a PCV lesion with the greatest linear dimension of <6 mm, but not greater than 3 mm from the center of the fovea to the furthest point on lesion perimeter (determined by ICG).
* The distance from the center of the fovea to the nearest edge of the optic disc should be not less than 3 mm. (This distance is confirmed by Oraya software prior to treatment.).
* Must have provided informed consent, documented it in writing, and have been given a copy of the signed informed consent form.
* Must be willing and able to return for scheduled visits for the 2-year duration of the study.
* Must be at least 50 years of age.
* Women must be post-menopausal ≥1 year or surgically sterilized, or a pregnancy screen must be performed prior to the study and a reliable form of contraception, approved by the investigator, must be maintained during the study.
* Must have best corrected visual acuity of 75 to 25 letters (inclusive) in the study eye and at least 20 letters in the fellow eye (if both eyes meet all the study criteria, then the eye with the worst vision should be selected as the study eye).

Exclusion Criteria:

* CNV due to causes other than AMD or PCV, including ocular histoplasmosis syndrome, angioid streaks, multifocal choroiditis, choroidal rupture, or pathologic myopia (spherical equivalent -8 diopters).
* A globe axial length of <20 mm or >26 mm.
* Evidence of diabetes or with retinal findings consistent with diabetic retinopathy or retinopathy for any other cause.
* Hypertension that is not controlled with anti-hypertensive medication.
* Prior or concurrent therapies for age related macular degeneration or PCV, including submacular surgery, subfoveal thermal laser photocoagulation (with or without photographic evidence), or transpupillary thermotherapy (TTT).
* History of radiation to the head in the region of the study eye.
* Previous posterior vitrectomy at any time, YAG capsulotomy or cataract surgery within 3 months, or any other surgery in the study eye within 6 months prior to the screening visit.
* Intravitreal device in the study eye.
* Concomitant disease in the study eye which might interfere with the effect of assessment of the study treatment, including uveitis, acute ocular or periocular infection, retinal vasculopathies (including retinal vein occlusions, etc.) or intraocular pressure >30 mmHg uncontrollable with medications.
* History of rhegmatogenous retina detachment, optic neuritis or intraocular tumors in the study eye.
* Inadequate pupillary dilation, significant media opacities, or other conditions in the study eye, including cataract, which may interfere with visual acuity or the evaluation of the posterior segment. Subjects likely to need cataract surgery during the 1 year study period should also not be enrolled.
* Known serious allergies to fluorescein or indocyanine green dye used in angiography.
* Subjects must not have subretinal hemorrhage or Retinal Pigment Epithelium tear involving the center of the foveal avascular zone.
* Known sensitivity or allergy to Lucentis, or any other drug used in the study, such as topical anesthetic, cycloplegic mydriatics, or lubricating eye gel.
* Contraindication or sensitivity to contact lens application (i.e. corneal dystrophies and recurrent corneal erosions). 16. Currently receiving chemotherapy, having completed a course within the 90 days preceding study enrollment, or expecting to begin chemotherapy while participating in the study.
* Current participation in another PCV drug or device clinical trial.
* History of use of drugs with known retinal toxicity, including: chloroquine (Aralen - antimalarial), hydroxychloriquine (Plaquenil - antimalarial), phenothiazines (Thorazine, Stelazine, Mellaril, Prolixin, Trilafon, etc., - tranquilizing antipsychotic medications) and these patients are exhibiting signs of retinal toxicity.
* Concurrent use of systemic anti-VEGF agents.
* Any other condition, which in the judgment of the investigator would prevent the subject from granting consent or completing the study, such as dementia, mental illness (including generalized anxiety disorder, claustrophobia, etc.), or inability to position in the device (due to musculoskeletal problems, etc.).
* History of other significant, uncontrolled disease including cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal, metabolic dysfunction, any clinical finding giving reasonable suspicion of a disease or condition that contraindicates the use of intravitreal ranibizumab or that might affect interpretation of the results of the study or render the subject at high risk for treatment complication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Lesion change as measured with fluorescein angiography. | Baseline and 12 months
  Change in the proportion of the lesion which is active at 12 months.

SECONDARY OUTCOMES:
Number of Lucentis injections | baseline and 12 months
  Number of Lucentis injections during 12 months
Visual Acuity change | Baseline and 12 months
  Mean change in visual acuity
Polyp changes | Baseline and 12 months
  Change in total lesion and polyp size & number of polyps

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita-Salute Istituto Scientifico San Raffaele, Milan, Italy